CLINICAL TRIAL: NCT02436278
Title: Does 4 Metre Gait Speed (4MGS) Predict Mortality and Non-elective Hospitalisation in Patients With Idiopathic Pulmonary Fibrosis (IPF)?
Brief Title: The Predictive Ability of 4MGS in IPF
Acronym: IPFMORT
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/LO/0015
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Gait speed; Mortality; Morbidity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPF_MORT: Patients diagnosed with Idiopathic Pulmonary Fibrosis according to NICE guidelines.
  Interventions: Other: 4MGS

INTERVENTIONS:
Other: 4MGS — Usual walking speed measured over 4 metres

SUMMARY:
This study investigates whether usual walking speed, measured by the 4 metre gait speed test (4MGS), and change in usual walking speed over 6 months predicts death and hospital admissions in patients with Idiopathic Pulmonary Fibrosis.

DETAILED DESCRIPTION:
This observational study is investigating a simple test of usual walking speed, measured using the 4 metre gait speed (4MGS) test in patients with a lung disease called Idiopathic Pulmonary Fibrosis (IPF). Drug development for this disease is slow in part because there is a lack of reliable measurements that can assess the effectiveness of treatment. Death and hospital admissions are currently considered meaningful endpoints in research trials due to the lack of fully validated surrogate endpoints in IPF. Using surrogate endpoints could reduce the sample size, cost and duration of clinical trials in IPF perhaps permitting more rapid drug development. Slow walking speed has been shown to be consistently associated with survival and a risk factor for disability, institutionalisation and hospitalisation in older adults and people with another lung disease called Chronic Obstructive Pulmonary Disease (COPD). We are interested to see whether usual walking speed and change in usual walking speed over 6 months predicts death and hospital admissions in IPF patients. This will help inform us of the potential use of 4MGS as a surrogate endpoint. To do this, participants who consent to taking part in the study will be timed walking at their usual walking speed over a distance of 4 metres (13.12 feet) at one time point and then six months later. Incidence of mortality and non-elective hospital admissions will be assessed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis according to NICE guidelines

Exclusion Criteria:

* Significant co-morbidities that would limit walking ability, exercise capacity or make exercise unsafe (e.g. unstable ischaemic heart disease, neuromuscular disease, severe hip/lower limb joint pain, peripheral vascular disease, lower limb amputation)
* Any patient whom the chief investigator feels it is unsafe to exercise (e.g. unstable cardiovascular disease)
* Any condition that precludes providing informed consent e.g. cognitive impairment or poor English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IPF according to NICE guidelines
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  IPF-specific and all-cause mortality

SECONDARY OUTCOMES:
Non-elective hospital admissions | 12 months
  IPF-specific and all-cause hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MC, PhD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Harefield, Middlesex, United Kingdom

REFERENCES:
- [Derived] Nolan CM, Delogu V, Maddocks M, Patel S, Barker RE, Jones SE, Kon SSC, Maher TM, Cullinan P, Man WD. Validity, responsiveness and minimum clinically important difference of the incremental shuttle walk in idiopathic pulmonary fibrosis: a prospective study. Thorax. 2017 Sep 7:thoraxjnl-2017-210589. doi: 10.1136/thoraxjnl-2017-210589. Online ahead of print. PMID 28883090